CLINICAL TRIAL: NCT06753578
Title: Effectiveness of an ACT-Based Cognitive Intervention on Quality of Life and Cognitive Function in Elderly Residents With MCI
Acronym: EACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ACT
Record Dates: First submitted 2024-11-08; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Acceptance and Commitment Therapy; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT (Experimental)
  Interventions: Behavioral: Acceptance and Commitment Therapy (ACT)
- Standard care (Active Comparator)
  Interventions: Behavioral: standard care

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy (ACT) — Acceptance and Commitment Therapy (ACT); Quality of Life (QOL); Mild Cognitive Impairment (MCI); cognitive function; elderly; psychological flexibility.
  Arms: ACT
Behavioral: standard care — standard care
  Arms: Standard care

SUMMARY:
This study investigates the effects of an Acceptance and Commitment Therapy (ACT)-based cognitive intervention on Quality of Life (QOL) and cognitive function among elderly residents with Mild Cognitive Impairment (MCI) in long-term care settings. The study assesses immediate and long-term impacts on cognitive function, psychological flexibility, social engagement, and overall well-being through structured ACT-based training.

DETAILED DESCRIPTION:
This clinical trial explores the impact of an Acceptance and Commitment Therapy (ACT)-based cognitive intervention on Quality of Life (QOL) and cognitive function in elderly residents with Mild Cognitive Impairment (MCI) living in long-term care facilities. The intervention aims to promote psychological flexibility, which is a core process in ACT, and enhance the residents' ability to engage in meaningful activities despite cognitive limitations.

Participants will engage in structured ACT-based training sessions that include mindfulness exercises, values clarification, and commitment strategies designed to improve cognitive engagement, reduce emotional distress, and foster greater social connection. The study measures both the immediate effects following the intervention and the long-term benefits at follow-up periods to evaluate sustained improvements in cognitive performance, psychological resilience, social involvement, and overall well-being.

By focusing on cognitive and emotional strategies, the intervention seeks to empower elderly residents to live more fulfilling and value-driven lives, even in the face of cognitive decline associated with MCI.

ELIGIBILITY:
Inclusion Criteria:

* Residents aged 65 and older diagnosed with MCI, able to provide informed consent, and residing in participating long-term care facilities.

Exclusion Criteria:

* Individuals with severe cognitive impairment, unstable medical conditions, or psychiatric diagnoses that would interfere with participation.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 215 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life as measured by the QOL-AD scale | Baseline, post-intervention (12 weeks), and 6-month follow-up
  Quality of Life will be assessed using the QOL-AD scale, a validated questionnaire for evaluating the quality of life in individuals with cognitive impairment. Changes in mean scores from baseline to each time point will be reported
Change in cognitive function as measured by the Mini-Mental State Examination (MMSE) | Baseline, post-intervention (12 weeks), and 6-month follow-up
  Cognitive function will be evaluated using the MMSE, a widely used tool for cognitive assessment. Mean changes in scores from baseline to each time point will be analysed and reported

SECONDARY OUTCOMES:
Psychological flexibility as measured by the Acceptance and Action Questionnaire (AAQ-II) | Baseline, post-intervention (12 weeks), and 6-month follow-up
  Psychological flexibility will be measured using the AAQ-II, a validated scale assessing an individual's ability to engage with values-based actions despite cognitive and emotional challenges. Mean score changes over time will be reported
Social engagement as measured by a standardised engagement assessment tool | Baseline, post-intervention (12 weeks), and 6-month follow-up
  Social engagement will be assessed using a standardised instrument for evaluating participation in meaningful activities and interpersonal connections. Changes in engagement levels will be tracked and reported

CONTACTS AND LOCATIONS:
Locations (1):
- Religious congregation, Santander, Cantabria, Spain

IPD SHARING:
Plan to Share IPD: No